CLINICAL TRIAL: NCT01897389
Title: A Single-Dose, Open-Label, Randomized, 4-Period, 5-Treatment Crossover Study to Assess the Relative Bioavailability of 4 New Abiraterone Acetate Tablet Formulations With Respect to the Current Commercial Abiraterone Acetate Tablet Under Fasted Conditions in Healthy Male Subjects
Brief Title: A Study to Assess the Relative Bioavailability of 4 New Abiraterone Acetate Tablet Formulations With Respect to the Current Commercial Abiraterone Acetate Tablet Under Fasted Conditions in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR102353; 212082PCR1010 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Bioavailability; Abiraterone acetate; ZYTIGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Sequence 1: abiraterone acetate (Experimental): Treatment sequence 1 is defined as: AEBD
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment D; Drug: Treatment E
- Sequence 2: abiraterone acetate (Experimental): Treatment sequence 2 is defined as: BACE
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment E
- Sequence 3: abiraterone acetate (Experimental): Treatment sequence 3 is defined as: CBDA
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D
- Sequence 4: abiraterone acetate (Experimental): Treatment sequence 4 is defined as: EDAC
  Interventions: Drug: Treatment A; Drug: Treatment C; Drug: Treatment D; Drug: Treatment E
- Sequence 5: abiraterone acetate (Experimental): Treatment sequence 5 is defined as: DECA
  Interventions: Drug: Treatment A; Drug: Treatment C; Drug: Treatment D; Drug: Treatment E
- Sequence 6: abiraterone acetate (Experimental): Treatment sequence 6 is defined as: EADB
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment D; Drug: Treatment E
- Sequence 7: abiraterone acetate (Experimental): Treatment sequence 7 is defined as: ABEC
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment E
- Sequence 8: abiraterone acetate (Experimental): Treatment sequence 8 is defined as: BCAD
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D

INTERVENTIONS:
Drug: Treatment A — 1000 mg abiraterone acetate (4 250-mg tablets - current commercial formulation, reference drug) administered as a single oral dose under fasted conditions
Drug: Treatment B — 1000 mg abiraterone acetate (4 250-mg tablets - new formulation) administered as a single oral dose under fasted conditions
  Arms: Sequence 1: abiraterone acetate; Sequence 2: abiraterone acetate; Sequence 3: abiraterone acetate; Sequence 6: abiraterone acetate; Sequence 7: abiraterone acetate; Sequence 8: abiraterone acetate
Drug: Treatment C — 1000 mg abiraterone acetate (2 500-mg tablets - new formulation) administered as a single oral dose under fasted conditions
  Arms: Sequence 2: abiraterone acetate; Sequence 3: abiraterone acetate; Sequence 4: abiraterone acetate; Sequence 5: abiraterone acetate; Sequence 7: abiraterone acetate; Sequence 8: abiraterone acetate
Drug: Treatment D — 1000 mg abiraterone acetate (4 250-mg tablets - same composition as current commercial formulation) administered as a single oral dose under fasted conditions
  Arms: Sequence 1: abiraterone acetate; Sequence 3: abiraterone acetate; Sequence 4: abiraterone acetate; Sequence 5: abiraterone acetate; Sequence 6: abiraterone acetate; Sequence 8: abiraterone acetate
Drug: Treatment E — 1000 mg abiraterone acetate (2 500-mg tablets - same composition as current commercial formulation) administered as a single oral dose under fasted conditions
  Arms: Sequence 1: abiraterone acetate; Sequence 2: abiraterone acetate; Sequence 4: abiraterone acetate; Sequence 5: abiraterone acetate; Sequence 6: abiraterone acetate; Sequence 7: abiraterone acetate

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of 4 new formulations of abiraterone acetate compared to the current commercial formulation.

DETAILED DESCRIPTION:
This is a randomized (individuals will be assigned by chance to study treatments), open-label (individuals will know the identity of study treatments), 4-period, 5-treatment crossover study in order to evaluate the relative bioavailability of 4 new formulations of abiraterone acetate compared to the current commercial formulation. Approximately 32 healthy adult males will participate. The total study length is up to 68 days. This study will consist of a screening phase followed by an open-label treatment phase consisting of 4 single-dose treatment periods separated by a washout period of at least 7 days between dosing. Individuals will be randomly assigned to 1 of 8 treatment sequences. A single dose of 1000 mg abiraterone acetate will be given in each treatment period under fasted conditions. Participants will be confined to the study center from Day -1 of each treatment period until completion of the 96-hour blood sample collection on Day 5 of each treatment period. A follow-up visit will occur between 5 to 7 days after the last study procedure. Serial pharmacokinetic (study of what the body does to a drug) samples will be collected during the open-label treatment phase as detailed in the protocol. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to protocol-defined use of effective contraception for up to 1 week after receiving the last dose of study drug and agrees to not donate sperm during the study and for 1 week after receiving the last dose of study drug
* Body mass index between 18.5 and 30.0 kg/m2 (inclusive) and body weight not less than 50 kg
* Blood pressure (after lying down for 5 minutes) between 90 and 140 mmHg systolic and no higher than 90 mmHg diastolic
* A 12-lead electrocardiogram consistent with normal cardiac conduction and function
* Non-smoker and no use of nicotine-containing substances within the previous 2 months
* Laboratory values within protocol-defined parameters

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the patient or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, urinalysis, or clinically significant abnormal physical examination, vital signs, or 12-lead electrocardiogram at screening or at admission to the study center as deemed appropriate by the investigator
* Screening serum testosterone level of <200 ng/dL
* Presence of sexual dysfunction or any medical condition that would affect sexual function
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, within 14 days before the first dose of the study drug is scheduled through study completion
* History of, or a reason to believe a participant has a history of drug or alcohol abuse within the past 5 years
* Positive test for drugs of abuse (such as cannabinoids, alcohol, opiates, cocaine, amphetamines, benzodiazepines, hallucinogens, or barbiturates) at screening and Day -1 of each treatment period
* Known allergy to the study drug or any of the excipients of the formulation
* History of stomach or intestinal surgery or resection that would potentially alter absorption or excretion of orally administered drugs (appendectomy and hernia repair will be allowed)
* Donated blood or blood products or had substantial loss of blood within 3 months before the first administration of study drug or intention to donate blood or blood products during the study
* Received an experimental drug or used an experimental medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before the first dose of the study drug is scheduled
* Unable to swallow solid, oral dosage forms whole with the aid of water
* Positive test for human immunodeficiency virus 1 and 2 antibodies, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibodies
* Preplanned surgery or procedures that would interfere with the conduct of the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of abiraterone | Periods 1-4 pharmacokinetic profile from Day 1 predose and postdose at 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h, 96 h
Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration of abiraterone | Periods 1-4 pharmacokinetic profile from Day 1 predose and postdose at 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h, 96 h
Area under the plasma concentration-time curve from time 0 to infinite time of abiraterone | Periods 1-4 pharmacokinetic profile from Day 1 predose and postdose at 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h, 96 h
Elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve of abiraterone | Periods 1-4 pharmacokinetic profile from Day 1 predose and postdose at 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h, 96 h
Time to reach the maximum plasma concentration of abiraterone | Periods 1-4 pharmacokinetic profile from Day 1 predose and postdose at 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h, 96 h

SECONDARY OUTCOMES:
Number of participants affected by adverse events by MedDRA system organ class (SOC) and Preferred term (PT) | Up to 30 days after the last dose of study medication

OTHER OUTCOMES:
Percentage of area under the plasma concentration-time curve from time 0 to infinite time obtained by extrapolation of abiraterone | Periods 1-4 pharmacokinetic profile from Day 1 predose and postdose at 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h, 96 h
First-order rate constant associated with the terminal portion of the drug-concentration-time curve of abiraterone | Periods 1-4 pharmacokinetic profile from Day 1 predose and postdose at 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h, 96 h
Time to last quantifiable plasma concentration of abiraterone | Periods 1-4 pharmacokinetic profile from Day 1 predose and postdose at 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h, 96 h

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States